CLINICAL TRIAL: NCT04194658
Title: The Effectiveness of Using Letrozole Prior to Misoprostol Versus Misoprostol Alone for Successful Induction of Medical Abortion: A Randomized Controlled Trial
Brief Title: Effectiveness of Pretreatment Letrozole Versus Misoprostol Alone in Missed Abortion
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Fathy Zaky, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Letrozole in missed abortion
Record Dates: First submitted 2019-12-09; First posted 2019-12-11 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Medical; Abortion, Fetus
MeSH Terms: interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case group (Active Comparator): Case group will receive pretreatment letrozole 12.5 mg for 2 days before administration of misoprostol in a dosage according to ACOG guidelines based on gestational age.
  Interventions: Drug: Letrozole 2.5mg
- Control group (No Intervention): Control group will receive only misoprostol in a dosage according to ACOG guidelines based on gestational age.

INTERVENTIONS:
Drug: Letrozole 2.5mg — Pretreatment letrozole 12.5 mg for 2 days prior to misoprostol.
  Arms: Case group

SUMMARY:
Background and Rationale Abortion accounts for about 8% of maternal mortality worldwide. Surgical intervention is the definitive treatment for abortion but it is invasive. Misoprostol, a PG E1 analogue, is exten¬sively used for induction of abortion with success rate less than 90%. Estrogen is important in the maintenance of pregnancy & aromatase enzyme is essential for its production. Letrozole is an aromatase inhibitor. So we assume that suppression of serum estradiol by letrozole will facilitate termination of pregnancy.

Objectives :

To compare the effect of a combination of letrozole with misoprostol versus misoprostol alone in successful induction of medical abortion.

Study population & Sample size 150 women will be recruited. Women included will be > 18 years with singleton pregnancy of gestational age ≤ 20 weeks having missed abortion. They will be excluded if they have prior CS, twin pregnancy, allergy to letrozole or liver problems.

Study Design :

A randomized controlled trial in which patients will be divided into 2 groups; case group & control group. Each group will contain 75 patients.

Methods :

Case group will receive pretreatment letrozole 12.5 mg for 2 days while control group will receive only misoprostol. Both groups will receive misoprostol in a dosage according to the ACOG guidelines based on gestational age.

Possible Risk (s) to study population :

Major risks (Sepsis, considerable vaginal bleeding leading to hemodynamic instability or necessitating blood transfusion). Minor risks (Nausea, diarrhea, headache, weakness, hot flushes).

Outcome parameter (s):

Successful medical abortion i.e. complete abortion with no need for surgical curettage within one week from the 1st dose of misoprostol.

DETAILED DESCRIPTION:
Background and Rationale:

Abortion management is one of the most important issues in gyne¬cology. According to the WHO abortion accounts for about 8% of maternal mortality worldwide. The term 'abortion' has become synonymous with induced abortion which is an intentional termination of pregnancy but it also includes spontaneous abortion.

Induced abortion is thus one of the most commonly investigated topics in gynecology as means to achieve safe abortion in order to reduce associated maternal morbidity & mortality.

Abortion is defined as the termination of a pregnancy before the 20th week of pregnancy or termina¬tion of pregnancy before the fetus weighing 500 g.

Surgical intervention is the definitive treatment for abortion. However, it is invasive and is not necessary for all females. Curettage may be avoided via expectation and medi¬cal treatment.

Misoprostol, a synthetic analogue of natural prostaglandin E1, is exten-sively used for early termination of pregnancy, therapeutic abortion, treatment of incomplete or missed abortion. It results in abortion by ripening of the cervix & stimulating the myometrium. Misoprostol abortion rate is less than 90% in most studies and it has different side effects.

Progesterone is an essential component to establish and maintain pregnancy. It is responsible for the transformation of the endometrium from a proliferative to a secretory state. In addition, it has a role in relaxation of the uterus and prevention of cervical dilatation.

Estrogen is also important in the maintenance of pregnancy, although less evidence exists for this. Aromatase enzyme is essential for its production via aromatization of androgens.

During early pregnancy, the corpus luteum is the main source of estrogen and progesterone. It is initially maintained by luteinizing hormone (LH) from the anterior pituitary, then after implantation human chorionic gonadotropin (hCG) from the trophoblastic cells takes over the role of LH. This continues until the 7th week of pregnancy, when the placenta becomes the main source of hormone production.

Pharmacological agents that can reduce or block the actions of progesterone or estrogen may therefore have a role in medical abortion.

Mifepristone, a progesterone antagonist, is widely used for medical abortion in countries where it is available. The complete abortion rate of the sequential regimen using 200 mg of oral mifepristone, followed 36-48 h later by a single dose of 800 µg of vaginal misoprostol, is over 95% in pregnancies of less than 9 weeks' gestation.

The widespread use of mifepristone is limited by the fact that it is expensive and not available in many countries. Therefore a cheaper and easily available alternative needs to be found.

Letrozole, a non-steroidal aromatase inhibitor, is most commonly used in hormone-sensitive breast cancer. It reversibly and competitively bonds with the iron in cytochrome P450 and prevents estrogen production by the enzyme aromatase.

Since estrogens are necessary for continuation of the pregnancy, we hypothesize that acute suppression of the serum estradiol concentration by letrozole in human pregnancy would affect the function of corpus and/or placenta thus facilitating termination of pregnancy.

Objectives:

To compare the effect of a combination of letrozole with misoprostol versus misoprostol alone in successful induction of medical abortion.

Study Design:

A randomized controlled trial involving 150 women will be performed. They will be randomly divided into 2 groups; each group contains 75 participants.

Case group will receive pretreatment letrozole 12.5 mg for 2 days while control group will receive only misoprostol. Both groups will receive misoprostol in a dosage according to the ACOG guidelines based on gestational age.

The study performed will be a phase 2 clinical trial. The study will be performed in Obstetrics & Gynecology Department, Kasr Al-Ainy Hospital, Cairo University.

Patient & Methods:

Sample size:

Sample size was calculated to prevent type II error. According to Naghshineh and coworkers (2015), complete abortion rates among case subjects was 76.7 % versus 42.6 % in the control subjects. Calculation showed we need 51women in each arm to be able to reject with a probability of 95% the null hypothesis that the rates for the case and control groups are equal. The type I error probability associated with this test for the null hypothesis was 0.05. Additionally, to compensate for subjects declining to participate or lost to follow-up, we recruited 75 women in each arm.

Statistical analysis The collected data will be tabulated and analyzed using appropriate statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy.
* Primigravida or multigravida.
* Gestational age ≤ 20 weeks.
* Missed abortion.

Exclusion Criteria:

* Maternal age < 18 years.
* Twin pregnancy.
* Previous cesarean section.
* Allergy to letrozole or misoprostol.
* Liver cirrhosis or severe liver impairment.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Successful medical abortion | One week from the 1st dose of misoprostol.
  Number of participants who achieved complete abortion with no need for surgical intervention in each group

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Seleem, MD, Study Director — Cairo University

REFERENCES:
- [Background] Yung SSF, Lee VCY, Chiu PCN, Li HWR, Ng EHY, Yeung WSB, Ho PC. The effect of 7 days of letrozole pretreatment combined with misoprostol on the expression of progesterone receptor and apoptotic factors of placental and decidual tissues from first-trimester abortion: a randomized controlled trial. Contraception. 2016 Apr;93(4):323-330. doi: 10.1016/j.contraception.2015.12.005. Epub 2015 Dec 19. PMID 26707996
- [Background] Naghshineh E, Allame Z, Farhat F. The effectiveness of using misoprostol with and without letrozole for successful medical abortion: A randomized placebo-controlled clinical trial. J Res Med Sci. 2015 Jun;20(6):585-9. doi: 10.4103/1735-1995.165964. PMID 26600834